CLINICAL TRIAL: NCT06218147
Title: Community-Based Nutrition-Lifestyle Therapy for Pregnant Latina Women With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sansum Diabetes Research Institute (Other)
Responsible Party: Principal Investigator, Rachyl Pines, Adjunct Research Scientist, Sansum Diabetes Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCON-00003510
Record Dates: First submitted 2023-12-22; First posted 2024-01-23 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Mel Gestational - in Pregnancy
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard care group (No Intervention): Participants in this group will meet with their CHW for 8 sessions (almost weekly from weeks 14 to 27 gestation) and then 4 sessions (almost biweekly from weeks 28-35 gestation) to match the contact provided in dietary-lifestyle behavioral intervention group. Sessions will be held in person, with videoconferencing and phone call options available when in person is not possible. In these brief check-in sessions, the CHW will be focused on maintaining regular contact, connecting participants to community resources, checking in about any new or ongoing medical issues described by participant during each session visit, and providing overall general information about diabetes management when indicated. CGM will be blinded for both groups.
- Nutrition-behavior lifestyle program group (Experimental): Participants in this group meet with their CHWs for 8 sessions (almost weekly from weeks 14 to 27 gestation) and then 4 sessions (almost biweekly from weeks 28-35 gestation). Sessions are held in person, with videoconferencing and phone call options available when in person is not possible. CGM wear is blinded in both groups. The topics for each session are:
  1. Welcome and Understanding Diabetes in Pregnancy
  2. Understanding Food Groups & Setting Goals
  3. Understanding Carbohydrate Types & Portions
  4. Reading Nutrition Labels & Understanding Added Sugar
  5. Exercise in Pregnancy & Carbohydrate Counting
  6. Grocery Shopping & Using SNAP or WIC Benefits
  7. Managing Stress - Communal Coping as a Family
  8. Getting Ready for Baby & My Family Plan
  9. How to Receive Social Support
  10. Making Choices at Restaurants & Social Eating Settings
  11. Learning Empowered Communication with Providers
  12. Maintaining Changes & Staying Motivated
  Interventions: Behavioral: Nutrition-behavior lifestyle program

INTERVENTIONS:
Behavioral: Nutrition-behavior lifestyle program — The 15 participants randomized to the intervention group will complete the activities described in the arm/group description.
  Other Names: Plant forward dietary lifestyle intervention
  Arms: Nutrition-behavior lifestyle program group

SUMMARY:
Socioeconomically disadvantaged (SED) pregnant Latina women are disproportionately burdened by type 2 diabetes (T2D). Although lifestyle interventions can help to improve diabetes control, there are barriers to SED, Spanish-speaking pregnant people participating. The purpose of this proposal is to develop and test a culturally tailored, dietary-lifestyle behavioral intervention that supports eating plant-based foods such as fruits, vegetables, nuts and grains instead of processed foods and meat, and is implemented through community health workers (CHWs) to prevent excessive weight gain during pregnancy and improve control of blood sugar levels in pregnant Latina women with T2D. This study takes advantage of our existing strong relationships with the local Latino community, CHWs, and Santa Barbara County Public Health, which includes eight multidisciplinary healthcare clinics with sliding fee programs, and Rooted Santa Barbara, a community plant-based lifestyle organization. Cultural sensitivity focuses on delivering health information based on norms, values, beliefs, environmental factors, and historical context that is unique to a racial/ethnic population. Therefore, for our program to be culturally sensitive, it will include delivery of the program by CHWs primarily in the Spanish language with English as needed and incorporation of culturally relevant eating and physical activity recommendations. The specific aims of the project are: 1) in year one, develop the dietary-lifestyle behavioral intervention that encourages a plant-forward diet for pregnant Latina women with T2D to prevent excessive weight gain during pregnancy and improve blood sugar control in collaboration with CHWs and participants by conducting focus groups to incorporate feedback on the program; 2) initiate in year one, and in year two, conduct a randomized controlled trial with 30 pregnant Latina women with T2D to evaluate the how well the nutrition-behavior lifestyle program works; and 3) evaluate the acceptance and delivery of the dietary-lifestyle behavioral intervention in CHWs and participants. If successful, this study will establish the how well a culturally sensitive program delivered by CHWs incorporating plant-forward diets for pregnant Latina women with T2D prevents excessive weight gain during pregnancy, and control of blood sugar levels.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes in pregnancy
* ≥ 18 years old
* Self-reported Hispanic and/or Latino/a heritage
* BMI ≥ 26.0 kg/m2 and ≤ 42.0 kg/m2

Exclusion Criteria:

* Type 1 Diabetes
* Active substance abuse with alcohol or drugs by self-report
* Treatment with non-diabetes medications (e.g., corticosteroids, anti-psychotics) known to have metabolic/body weight effects that could affect outcome measures
* Non-singleton fetus
* Evidence of fetal malformation
* HbA1c ≥ 10%
* Unable to provide informed consent or unwilling to complete the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
Percent of glucose time in range assessed by using continuous glucose monitor | 30 days at baseline and at 27 weeks gestation, and at 35 weeks gestation.
  All participants will wear a Continuous Glucose Monitor for 30 days at three time points

SECONDARY OUTCOMES:
Amount of Gestational Weight Gain | assessed at baseline and post-intervention (approximately 27-35 weeks gestation)
  weight gain in kilograms by measurements on a scale during study visits
Change in Blood Pressure | assessed at baseline and post intervention (approximately 27-35 weeks gestation)
  systolic and diastolic blood pressure
Amount of satisfaction with the Intervention | evaluated immediately post-intervention
  self-reported satisfaction satisfaction with the intervention assessed by surveys created for the purposes of this study

CONTACTS AND LOCATIONS:
Overall Officials: Rachyl Pines, PhD, Principal Investigator — Sansum Diabetes Research Insititute
Locations (1):
- Sansum Diabetes Research Institute, Santa Barbara, California, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared